CLINICAL TRIAL: NCT01265667
Title: A Phase 2/3 Randomized, Double-Blind, Placebo-Controlled, Dose-Finding Study of the Efficacy and Safety of Daily CF101 Administered Orally in Patients With Moderate-to-Severe Plaque Psoriasis
Brief Title: Trial of CF101 to Treat Patients With Psoriasis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Can-Fite BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CF101-202PS
Record Dates: First submitted 2010-12-09; First posted 2010-12-23 (Estimated); Results first posted 2017-09-20 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-10

CONDITIONS: Plaque Psoriasis
Keywords: Psoriasis; Plaque psoriasis
MeSH Terms: conditions — Psoriasis | interventions — CF101; N(6)-(3-iodobenzyl)-5'-N-methylcarboxamidoadenosine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CF101 2 mg (Experimental): CF101 2mg oral tablets
  Interventions: Drug: CF101
- Placebo (Placebo Comparator): Placebo oral tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CF101 — orally q12h
  Other Names: IB-MECA
  Arms: CF101 2 mg
Drug: Placebo — orally q12h
  Other Names: Dummy pills
  Arms: Placebo

SUMMARY:
Eligible patients with Psoriasis will be treated with CF101 or placebo twice daily for 16 weeks. All subjects will receive open-lable CF101 in weeks 17-32.

DETAILED DESCRIPTION:
Eligible patients will be randomly assigned to parallel dosing groups of CF101 2 mg or matching placebo tablets twice daily (BID) in a 1:1 ratio for the 16-week controlled treatment period. Approximately 94 patients will be assigned to each group.

Medication will be taken orally BID for 16 weeks in a double-blinded fashion. At the end of 16 weeks, all patients assigned to CF101 will continue CF101, while patients originally assigned to placebo will be reassigned to CF101.

Assessment of peripheral blood mononuclear cell (PBMC) adenosine A3 receptor (A3AR) expression at baseline and during treatment with CF101 in selected sites.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 80 years of age, inclusive
* Diagnosis of moderate-to-severe chronic plaque-type psoriasis with body surface area involvement ≥10%
* Duration of psoriasis of at least 6 months
* Physician global assessment (PGA) ≥3
* Candidate for systemic treatment or phototherapy for psoriasis
* Electrocardiogram (ECG) is normal
* Females of child-bearing potential must have a negative serum pregnancy test
* Females of child-bearing potential must be willing to use 2 methods of contraception
* Ability to complete the study in compliance with the protocol
* Ability to understand and provide written informed consent.

Exclusion Criteria:

* Erythrodermic, guttate, palmar, plantar, or generalized pustular psoriasis
* Treatment with systemic retinoids, corticosteroids, or immunosuppressive agents within 4 weeks of the Baseline visit
* Treatment with high potency topical corticosteroids, keratolytics, or coal tar within 2 weeks of the Baseline visit
* Ultraviolet or Dead Sea therapy within 4 weeks of the Baseline visit
* Treatment with a biological agent within a period of time equal to 5 times its circulating half-life
* Treatment with lithium, hydroxychloroquine or chloroquine within 2 weeks of the Baseline visit
* Serum creatinine level greater than 1.5 times the laboratory's upper limit of normal
* Liver aminotransferase levels greater than the laboratory's upper limit of normal
* Significant acute or chronic medical or psychiatric illness
* Participation in another investigational drug or vaccine trial concurrently or within 30 days prior to Screening visit.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 293 (Actual)
Dates: Start 2011-07; Primary Completion 2015-03 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Silverman, MD, Study Director — Can-Fite BioPharma
Locations (18):
- Mount Sinai School of Medicine, New York, New York, United States
- Bulgaria (8):
  - UMHAT "G.stranski", Pleven
  - MHAT "Tokuda hospital Sofia", Sofia
  - DCC "Fokus-5"-MIOC, EOOD, Sofia
  - Military Medical Acdemy (MMA), Sofia
  - MHAT "Doverie", Sofia
  - City Center for Skin and Venereal Disease, Sofia
  - Multiprofile Hospital for Active Ttreatment, Stara Zagora
  - MHAT Varna at MMA Sofia, Varna
- Israel (3):
  - Haemek Medical Center, Afula
  - Rambam Medical Center, Haifa
  - Rabin Medical Center, Petah Tikva
- Romania (6):
  - Centrul Medical Euromed, Bucharest
  - Spitalul Clinic Dermato-Venerice, Bucharest
  - Emergency County Clinical Hospital, Cluj-Napoca
  - Spitalul Clinic Judetean de Urgenta Constanta, Constanța
  - Spit Clinic Judetean de Urgenta Sf Spiridon Iasi, Iași
  - County Clinical Emergency Hospital, Sibiu

REFERENCES:
- See also: Can-Fite BioPharma website — http://www.canfite.com/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CF101 2 mg | Placebo
Started | 145 | 148
Completed | 125 | 135
Not Completed | 20 | 13

BASELINE CHARACTERISTICS:
Groups:
- CF101 2mg; Placebo: Oral tablets given every 12 hours for 16 weeks
- Total: Total of all reporting groups
Arm/Group | CF101 2mg | Placebo | Total
Number analyzed (Participants) | 145 | 148 | 293
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.3 (13.57) | 50.0 (13.96) | 49.2 (13.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 53 | 107
  Male | 91 | 95 | 186

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Achieving Psoriasis Area and Severity Index (PASI) 75 at 12 Weeks
Description: Achievement of PASI 75 indicates a 75% reduction in the PASI score, which ranges from 0 (no disease) to 72 (maximal disease)
Time Frame: 12 weeks
Population: Analysis was performed on the Intent-to-treat (ITT) Population
Measure: Count of Participants; unit: Participants
Arm/Group | CF101 2 mg | Placebo
Number analyzed (Participants) | 141 | 144
Participants | 12 | 10

2. Secondary Outcome: Number of Subjects Achieving PGA of 0 or 1
Description: PGA is a physician's assessment of the severity of disease based on a 6-point scale (score of 0 = clear and 5 = very severe)
Time Frame: 16 weeks
Population: Analysis was performed on the ITT population
Measure: Number; unit: participants
Arm/Group | CF101 2 mg | Placebo
Number analyzed (Participants) | 141 | 144
participants | 9 | 5

3. Secondary Outcome: Numberof Patients Achieving Psoriasis Area and Severity (PASI) Score of 50 or 75
Description: Achievement of PASI 50 or 75 indicates a 50% and 75% reduction respectively in the PASI score, which ranges from 0 (no disease) to 72 (maximal disease)
Time Frame: 16 weeks
Population: Analysis performed of the ITT population
Measure: Number; unit: participants
Arm/Group | CF101 2 mg | Placebo
Number analyzed (Participants) | 141 | 144
participants | 31 | 17

4. Secondary Outcome: Nature and Frequency of Adverse Events
Description: Assessment of safety of CF101 in this patient population by gathering adverse event data based on history, vital signs, physical examination, and laboratory data
Time Frame: 32 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | CF101 2 mg | Placebo
Number analyzed (Participants) | 145 | 148
Participants
  Any | 37 | 29
  Gastrointestinal disorders | 8 | 3
  Infections and infestations | 10 | 13
  Musculoskeletal and connective tissue disorders | 5 | 2
  Nervous system disorders | 6 | 0
  Renal and urinary disorders | 5 | 4

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: All adverse events were collected and verbatim terms were coded via MedDRA dictionary
Arm/Group | CF101 2 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/145 | 0/148
Other Adverse Events (participants affected / at risk) | 24/145 | 15/148
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CF101 2 mg (N=145) | Placebo (N=148)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Influenza (Infections and infestations) | 0 | 2
Nasopharyngitis (Infections and infestations) | 2 | 2
Urinary tract infection (Infections and infestations) | 2 | 4
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Dry mouth (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 2
Headache (Nervous system disorders) | 4 | 0
Haematuria (Renal and urinary disorders) | 2 | 2
Proteinuria (Renal and urinary disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No